CLINICAL TRIAL: NCT06851351
Title: Study of Respiratory Restriction in Patients With Prader-Willi Syndrome
Brief Title: Respiratory Restriction in Prader-Willi Syndrome
Acronym: RESPIPWS
Status: Completed | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 01C318
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Prader-Willi Syndrome
Keywords: thoraco-abdominal volumes; lung volumes; optoelectronic plethysmography; respiratory manoeuvres; posture
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Spirometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Prader Will syndrome and BMI > 30 kg/m2
  Interventions: Diagnostic Test: Spirometry and optoelectronic plethysmography
- Control subjects with BMI < 25 kg/m2
  Interventions: Diagnostic Test: Spirometry and optoelectronic plethysmography

INTERVENTIONS:
Diagnostic Test: Spirometry and optoelectronic plethysmography — Spirometry for respiratory function and optoelectronic plethysmography for respiratory pattern during wakefulness

SUMMARY:
The main aim of this study is therefore to evaluate the impact of Prader Willi Syndrome (PWS) on lung and thoracoabdominal volumes, respiratory muscle strength and awake ventilatory pattern, and to quantify and localize the PWS-induced respiratory restriction.

DETAILED DESCRIPTION:
The aim is to study lung function in obese PWS patients using both volitional (spirometry, nitrogen wash-out, and maximal pressure measurements (MIP and MEP)) and non-volitional (awake ventilatory pattern by opto-electron plethysmography) tests, both in sitting and supine positions.

Spirometry, nitrogen wash-out, and MIP and MEP measurements are comprehensive assessments, while optoelectronic plethysmography allows restriction location through accurate measurement of thoracoabdominal volumes.

The results of the study could provide useful information about the calculation of the volumes enclosed by the grid of markers (in particular, the volume of the rib cage, which reflects the action of the intercostal muscles, the volume of the abdomen, which reflects the action of the diaphragm in the inspiratory phase and of the abdominal muscles during exhalation and their sum, which represents the total variation of the thoraco-abdominal wall. All these finds could be useful for respiratory rehabilitation protocols for obese PWS patients.

ELIGIBILITY:
Patients with Prader Willi Syndrome

Inclusion Criteria:

* Age 20-50 years
* Prader Willi Syndrome
* Body Mass Index > 30 kg/m2

Exclusion Criteria:

* Lack of signed consent form

Control subjects

Inclusion Criteria:

* Age 20-50 years
* Body Mass Index < 25 kg/m2

Exclusion Criteria:

* Lack of signed consent form

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Prader Willi Syndrome and obesity
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Rib cage contribution to ventilation | At enrollment
  Percentage rib cage contribution to ventilation as measured by optoelectronic plethysmography

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Site Piancavallo, Oggebbio, Verbania, Italy